CLINICAL TRIAL: NCT04353492
Title: A Single-arm, Prospective, Multicentre, Open-label Study to Evaluate Ofatumumab Treatment Effectiveness and Patient-reported Outcomes (PRO) in Patients With Relapsing Multiple Sclerosis (RMS) Transitioning From Fumarate-based RMS Approved Therapies or Fingolimod
Brief Title: An Open-label Study Evaluating Ofatumumab Treatment Effectiveness and PROs in Subjects With RMS Transitioning From Fumarate-based RMS Approved Therapies or Fingolimod to Ofatumumab
Acronym: ARTIOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMB157G23101; 2019-001341-40 (EudraCT Number)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: RMS; MS; multiple sclerosis; relapsing multiple sclerosis; OMB157; adult; secondary progressive MS; SPMS
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): Ofatumumab 20 mg subcutaneous injections every 4 weeks, following loading of 3 doses in the first 14 days
  Interventions: Biological: Ofatumumab

INTERVENTIONS:
Biological: Ofatumumab — Subjects will receive ofatumumab injections in an autoinjector (AI) for subcutaneous administration containing 20 mg ofatumumab (50 mg/ml, 0.4 ml content)
  Other Names: OMB157

SUMMARY:
Open-label study to evaluate the effectiveness of treatment with ofatumumab in subjects transitioning from any fumarate-based RMS approved therapy or fingolimod due to breakthrough disease.

DETAILED DESCRIPTION:
This was a single arm, prospective, multicentre and open-label, 96-week study to evaluate the treatment effectiveness of ofatumumab (OMB) in subjects with relapsing multiple sclerosis (RMS) transitioning from fumarate-based RMS approved therapies, such as dimethyl fumarate (DMF), diroximel fumarate (DRF), and monomethyl fumarate (MMF), or fingolimod due to breakthrough disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to the 2017 Revised McDonald criteria
* Relapsing MS: relapsing forms of MS (RMS) including RMS and secondary progressive MS (SPMS)
* Disability status at screening defined by Expanded Disability Status Scale (EDSS) score of 0 to 4 (inclusive)
* MS treatment history with a maximum of 3 Disease Modifying Therapies (DMTs), where all fumarates are considered as one DMT
* Subject transitioning from either any fumarate-based RMS approved therapies, such as dimethyl fumarate (DMF) or diroximel fumarate (DRF), or fingolimod which was administered for a period of at least 6 months, as their last DMT before first study drug administration
* Breakthrough disease activity while the participant was adequately using fumarates or fingolimod prior to transitioning for a minimum of 6 months as evidenced by one or more clinically reported relapses or one or more signs of Magnetic Resonance Imaging (MRI) activity (e.g. Gd+ enhancement, new or enlarging T2 lesions)
* Neurologically stable within one month prior to first study drug administration

Exclusion Criteria:

* Subjects with primary progressive MS or SPMS without disease activity
* Subjects meeting criteria for neuromyelitis optica
* Disease duration of more than 10 years since diagnosis
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they are using highly effective forms of contraception during dosing and for at least 6 months after stopping study medication
* Subjects with active chronic disease of the immune system other than MS or with immunodeficiency syndrome
* Subjects with active systemic bacterial, fungal or viral infections (such as hepatitis, HIV, COVID-19), or known to have Acquired Immunodeficiency Syndrome (AIDS)
* Subjects with neurological symptoms consistent with Progressive Multifocal Leukoencephalopathy (PML) or with confirmed PML
* Subjects at risk of developing or having reactivation of syphilis or tuberculosis (e.g. subjects with known exposure to, or history of syphilis, or active or latent tuberculosis, even if previously treated), as confirmed by medical history or per local practice
* Subjects with active hepatitis B and C disease, assessed locally
* Have received any live or live-attenuated vaccines within 4 weeks prior to first study drug administration
* Have been treated with medications as specified or within timeframes specified (e.g. corticosteroids, ofatumumab, rituximab, ocrelizumab, alemtuzumab, natalizumab, daclizumab, cyclophosphamide, teriflunomide etc.)
* Subjects suspected of not being able or willing to cooperate or comply with study protocol requirements in the opinion of the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 562 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2025-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (111):
- United States (25):
  - Fullerton Neuro and Headache Ctr, Fullerton, California
  - CU Anschutz Med Campus, Aurora, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Memorial Healthcare System, Hollywood, Florida
  - Homestead Assoc In Research Inc, Homestead, Florida
  - Neurology Associates PA, Maitland, Florida
  - UM Department Of Neurology, Miami, Florida
  - Negroski Neurology, Sarasota, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University Of South Florida, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - Georgia Neurology and Sleep Medicine Assoc, Suwanee, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Cleveland Clinic Foundation, Las Vegas, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - Five Towns Neuroscience Research, Woodmere, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Neuroscience, Westerville, Ohio
  - Multiple Sclerosis Center of Excellence of OMRF, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Saturn Research Solutions LLC, Plano, Texas
  - INOVA Medical Group, Fairfax, Virginia
  - Ascension St Francis Center, Milwaukee, Wisconsin
- Argentina (3):
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán
- Australia (3):
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Parkville, Victoria
- Austria (4):
  - Novartis Investigative Site, Linz, Upper Austria
  - Novartis Investigative Site, Vienna, Vienna
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
- Bulgaria (4):
  - Novartis Investigative Site, Pleven, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Novartis Investigative Site, Toronto, Ontario, Canada
- Czechia (5):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Havířov
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Teplice
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Germany (11):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Cottbus, Brandenburg
  - Novartis Investigative Site, Osnabrück, Lower Saxony
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Westerstede Olden
- Greece (2):
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Thessaloniki
- Hungary (3):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Pécs
- Italy (4):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
- Latvia (2):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Riga
- Novartis Investigative Site, Beirut, Lebanon
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Morelia, Michoacán
- Novartis Investigative Site, Oslo, Norway
- Poland (5):
  - Novartis Investigative Site, Bydgoszcz, Woj Kujawsko Pomorskie
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Wroclaw
- Portugal (4):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Loures
  - Novartis Investigative Site, Porto
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Saudi Arabia (2):
  - Novartis Investigative Site, Riyadh, SAU
  - Novartis Investigative Site, Jeddah
- Slovakia (5):
  - Novartis Investigative Site, Banská Bystrica, Slovakia
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Nitra, Slovakia
  - Novartis Investigative Site, Trnava, Slovakia
- Slovenia (2):
  - Novartis Investigative Site, Maribor, Slovenia
  - Novartis Investigative Site, Ljubljana
- Spain (7):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Santa Cruz, Santa Cruz de Tenerife
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Basel, Switzerland
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Trabzon, Ortahisar
  - Novartis Investigative Site, Istanbul, Sancaktepe
  - Novartis Investigative Site, Izmir
- United Kingdom (2):
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 27 countries.
Pre-assignment Details: 666 subjects were screened and 562 subjects were enrolled. Study had an up to 60 days screening period including baseline.
Period: Overall Study
Arm/Group | Ofatumumab
Started | 562
Completed | 523
Not Completed | 39
Not completed — Subject decision | 24
Not completed — Physician Decision | 5
Not completed — Adverse Event | 3
Not completed — Pregnancy | 3
Not completed — Lost to Follow-up | 2
Not completed — Protocol deviation | 1
Not completed — Technical problems | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab
Number analyzed (Participants) | 562
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.65)
Age, Customized [Count of Participants; unit: Participants]
  18 to 30 years | 185
  31 to 40 years | 181
  41 to 55 years | 190
  >55 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 369
  Male | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68
  Not Hispanic or Latino | 480
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 550
  More than one race | 0
  Unknown or Not Reported | 0
Number of relapses in the last 12 months prior to screening [Mean (Standard Deviation); unit: relapses] | 0.9 (0.71)
Number of relapses in the last 12 to 24 months prior to screening [Mean (Standard Deviation); unit: relapses] | 0.8 (1.04)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR)
Description: ARR is the number of confirmed relapses in a year calculated based on cumulative number of relapses by patient (adjusted for time-in-study by patient). Confirmed relapses are those accompanied by a clinically relevant change in the expanded disability status scale (EDSS).
  ARR was estimated from fitting a negative binomial regression model with log-link, and adjusted for prior MS therapies as a factor, number of relapses in previous year, baseline EDSS, baseline number of T1 Gd-enhancing lesions and the subject's age at baseline as covariates.
  The primary analysis describes the ARR with one-sided 95% confidence bound and test for null hypothesis (H0): ARR >=0.18 versus alternative hypothesis (H1): ARR<0.18.
Time Frame: Up to 96 weeks from baseline
Population: The Full Analysis Set (FAS) comprises all subjects to whom study treatment has been assigned and who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: relapses/ participant-year
Arm/Group | Ofatumumab
Number analyzed (Participants) | 562
relapses/ participant-year | 0.06 [0.05 to 0.08]
Statistical Analysis 1: Comparison: Ofatumumab; The null hypothesis (H0): ARR >= 0.18; Test type: Other — tested by a lower tailed test at 0.05 significance level; p < 0.0001, negative binomial regresion

2. Secondary Outcome: Number of of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of of participants with treatment emergent AEs and SAEs including injection related reactions, abnormal laboratory results or vital signs reported and qualifying as AEs.
Time Frame: From treatment day 1 to 100 days after last treatment up to approximatelly 26.6 months
Population: The Safety Set (SAF) includes all subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 562
Participants
  Adverse Events (AEs) | 509
  Serious Adverse Events (SAEs) | 33
  Treatment related AEs | 374
  AE causing study treatment discontinuation | 5
  AE causing study treatment interruption | 33

ADVERSE EVENTS:
Time Frame: From first dose of study treatment until 6 months after last dose up to 29.4 months approximately.
Groups:
- OMB 20mg: Ofatumumab 20 mg subcutaneous injections every 4 weeks, following loading of 3 doses in the first 14 days
Arm/Group | OMB 20mg
All-Cause Mortality (participants affected / at risk) | 0/562
Serious Adverse Events (participants affected / at risk) | 34/562
Other Adverse Events (participants affected / at risk) | 466/562
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg (N=562)
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Abscess limb (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Magnetic resonance imaging abnormal (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Medullary carcinoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebrovascular disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Multiple sclerosis relapse (Nervous system disorders) | 2
Optic neuritis (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Ureterolithiasis (Renal and urinary disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 1
Ovarian haematoma (Reproductive system and breast disorders) | 1
Ascites (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg (N=562)
Fatigue (General disorders and administration site conditions) | 34
Injection site reaction (General disorders and administration site conditions) | 62
COVID-19 (Infections and infestations) | 208
Influenza (Infections and infestations) | 29
Nasopharyngitis (Infections and infestations) | 96
Upper respiratory tract infection (Infections and infestations) | 78
Urinary tract infection (Infections and infestations) | 59
Injection related reaction (Injury, poisoning and procedural complications) | 300
Arthralgia (Musculoskeletal and connective tissue disorders) | 40
Back pain (Musculoskeletal and connective tissue disorders) | 40
Headache (Nervous system disorders) | 91
Cough (Respiratory, thoracic and mediastinal disorders) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT04353492/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT04353492/SAP_002.pdf